CLINICAL TRIAL: NCT06538571
Title: Association of Renal Near Infrared Spectroscopy in Outpatients With Parallel Circulation During the Interstage Period and Interstage Morbidity
Brief Title: Association of Near Infrared Spectroscopy With Interstage Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advocate Hospital System (Other)
Responsible Party: Principal Investigator, Joshua Wong, Principal Investigator, Advocate Hospital System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00111841
Record Dates: First submitted 2024-07-30; First posted 2024-08-05 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Single-ventricle
MeSH Terms: conditions — Univentricular Heart | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NIRS use (Experimental): Patients will have renal near infrared spectroscopy recorded in clinic.
  Interventions: Diagnostic Test: Near infrared spectroscopy

INTERVENTIONS:
Diagnostic Test: Near infrared spectroscopy — Noninvasive monitor for venous saturation

SUMMARY:
The purpose of this study is to assess the utility of renal near infrared spectroscopy in the outpatient setting during the interstage period. The primary aim will be to determine the correlation between oxygen extraction ratio ((arterial pulse oximetry - renal near infrared spectroscopy value)/arterial pulse oximetry value) with need for inpatient admission or intervention. Secondary aims will be to determine the correlation of the oxygen extraction ratio with weight gain, neurodevelopment, unexpected admissions, systemic ventricular strain by echocardiography, and Glenn hospitalization admission characteristics.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Infants under 6 months of age
* Infants with single ventricle heart disease and parallel circulation
* Infants who are awaiting the Glenn operation
* Infants who are outpatient

Exclusion Criteria:

* Infants over 6 months of age
* Inpatients
* Infants with history of skin injury from the near infrared spectroscopy sensor inpatient
* Infants with ongoing hyperbilirubinemia

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Unexpected admissions | 1 year
  The investigators will investigate the correlation between renal near infrared spectroscopy values and unexpected admissions during the interstage period.
Unexpected interventions | 1 year
  The investigators will investigate the correlation between renal near infrared spectroscopy values and unexpected need for interventions such as cardiac catheterization interventions or surgical interventions

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Wong, MD, Principal Investigator — Advocate Children's Hospital
Locations (1):
- Advocate Childrens Hospital, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No